CLINICAL TRIAL: NCT02259478
Title: Elucidation of the Mechanism of IVIG-Associated Hemolysis
Brief Title: Isoagglutinins in the Development of IVIG-associated Hemolysis
Status: Completed | Type: Observational
Sponsor: Toronto Transfusion Medicine Collaborative (Other)
Collaborators: University Health Network, Toronto (Other); Sunnybrook Health Sciences Centre (Other); Mount Sinai Hospital, New York (Other); The Hospital for Sick Children (Other); Unity Health Toronto (Other); Women's College Hospital (Other)
Responsible Party: Principal Investigator, Jacob Pendergrast, Consultant in Transfusion Medicine, Toronto Transfusion Medicine Collaborative
Other Study IDs: 14-8191-CE
Record Dates: First submitted 2014-08-29; First posted 2014-10-08 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Immunoglobulins, Intravenous; Hemolysis
Keywords: Intravenous Immunoglobulin (IVIG); Hemolysis; Transfusion Medicine; Pharmacovigilance
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected immediately prior and following a course of IVIG therapy, and then again 5-10 days later
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients at high risk of IVIG-associated hemolysis (defined as receipt of a 28-day cumulative dose of ≥ 2 g/kg, adjusted for ideal body weight, and non-O blood group) will be prospectively monitored using a standardized protocol for signs of hemolysis, and will be undergo additional testing for variables that have been hypothesized to increase the risk of hemolysis. The goal of the study is to define the incidence and dynamics of IVIG-mediated hemolysis and identify patient and product-related factors that may predict which patients are especially at risk.

DETAILED DESCRIPTION:
All IVIG orders received by the blood transfusion service at participating sites will be screened for patient eligibility. All non-O blood group patients receiving a cumulative 28-day dose of IVIG ≥ 2 g/kg will be approached for enrolment. Exclusion criteria include the presence of an alternate cause of anemia, including blood loss, other drug-induced hemolysis, anemia associated with chemotherapy for cancer, or hemolysis associated with an underlying disease or participation in another ongoing study. Patients receiving repeated courses of therapy will be eligible for re-enrollment a maximum of 6 times. There are otherwise no exclusions on the basis of age, diagnosis, concurrent treatment, or specific brand of product received. Enrolment will occur at multiple Canadian health care facilities.

Upon enrolment,case report forms documenting the participant's previous medical history, IVIG treatments and adverse reactions, and concurrent medication use will be collected. Laboratory testing for hemolysis will be performed at baseline, immediately following the completed high-dose cycle (usually administered over 1-2 days), and then again at 5-10 days post-infusion. IVIG associated. Hemolysis will be defined and graded as per the criteria of the Canadian IVIG Pharmacovigilance Group. The pathophysiology of IVIG-associated hemolysis will be characterized by tracking changes in serum complement levels, performing extended cytokine profiling, and conducting mononuclear phagocyte activity assays using patient monocytes. Secretor gene status, ABO zygosity and FcR polymorphisms will also be determined. A predictive model incorporating both patient factors (eg., blood group, total dose prescribed, presence of pre-infusion inflammation) and product factors (eg., specific lot number) will then be developed.

ELIGIBILITY:
Inclusion Criteria:

* cumulative dose within a 28-day period equal or greater to 2 g/kg body weight, adjusted for lean body mass
* non-O blood group
* willing to provide blood samples immediately prior to, immediately after the completion of, and 5-10 days after the course of IVIG therapy
* Able to provide informed consent, either themselves or through a surrogate decision-maker

Exclusion Criteria:

* evidence of active bleeding or hemolytic anemia at time of enrolment (patients with chronic, stable anemia will be eligible following review by the principle investigator)
* concurrently prescribed transfusion therapy

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All orders for IVIG received by the UHN Blood Transfusion Service will be reviewed by the study coordinator to identify potential study participants
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Hemolysis | From initiation of IVIG therapy to 5-10 days after the completion of last IVIG infusion
  Definition and grading of hemolysis adopted from the Canadian IVIG Hemolysis Pharmacovigilance Group

SECONDARY OUTCOMES:
Adverse transfusion reaction | From initiation of IVIG therapy to 5-10 days after the completion of last IVIG infusion
  Any patient symptom reported during or within 10 days of an IVIG infusion will be considered as a possible adverse transfusion reaction. Symptoms deemed to most likely indicate an adverse reaction include the development of fever, chills or rigours; allergic reactions (urticaria, angioedema or anaphylaxis); pain reactions (including headache); respiratory symptoms (cough, shortness of breath); and signs suggestive of anemia or hemolysis (pallor, fatigue, red-coloured urine, jaundice)
Descriptive analysis of risk factors | From initiation of IVIG therapy to 5-10 days after the completion of last IVIG infusion
  Additional secondary outcomes will include a descriptive analysis of information collected on the initial case report form such as patient demographics, medical history, dose and lot of IVIG administered, infusion rate, patient blood group, and concurrent medications. In addition, patient samples will be sent for additional testing aimed at elucidating the mechanism of IVIG-mediated hemolysis. These include:
  1. Cytokine panel profiling
  2. C3, C4, ferritin and CRP levels
  3. Monocyte monolayer assay using patient monocytes and implicated lot of IVIG against AET-treated group A1, B, and O red cells
  4. Tests of eluted IgG antibody for subtype.
  5. ABO zygosity (PCR) and/or by Flow
  6. FcR polymorphisms by PCR
  7. Secretor status by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Don Branch, PhD, Principal Investigator — Canadian Blood Services
Locations (6):
- Canada (6):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes